CLINICAL TRIAL: NCT02502071
Title: Effect of Urinary Alkalinization on Urine Uric Acid Precipitation and Crystallization in Adults With Type 1 DiabetesL a Open-label Trial
Brief Title: Effect of Urinary Alkalinization on Urine Uric Acid Precipitation and Crystallization in Adults With Type 1 Diabetes
Acronym: Alk-UA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-0541
Record Dates: First submitted 2015-07-16; First posted 2015-07-20 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Type 1 Diabetes; Diabetic Nephropathy; Diabetic Kidney Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Nephropathies | interventions — Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sodium Bicarbonate (Experimental): All participants will receive 2 doses of 1950mg Sodium Bicarbonate
  Interventions: Drug: sodium bicarbonate

INTERVENTIONS:
Drug: sodium bicarbonate — All participants will receive 2 doses of 1950mg sodium bicarbonate
  Other Names: NaHCO3

SUMMARY:
The purpose of this study is to determine whether alkalinization of urine uric acid by 2 doses of sodium bicarbonate (1950mg) over 24-hours reduces precipitation and crystallization of urine uric acid over in adults with type 1 diabetes.

DETAILED DESCRIPTION:
Diabetic nephropathy is characterized not only by glomerular disease but also tubulointerstitial injury. The tubular changes associated with diabetic nephropathy, include basement membrane thickening, tubular hypertrophy, epithelial-mesenchymal transition, glycogen accumulation and interstitial inflammation. Although glomerular changes has received significantly more attention from researchers and clinicians than tubulointerstitial changes in diabetes, tubular injury is known to associate better with renal function than glomerular injury. In fact, tubular proteinuria may precede microalbuminuria with type 1 diabetes, suggesting that tubular damage may be induced earlier than glomerular injury in the course of diabetic nephropathy.

Serum uric acid (SUA) is lower in adolescents and adults with type 1 diabetes compared to non-diabetic peers. Despite lower levels SUA remains an important risk factor for diabetic nephropathy in type 1 diabetes, with a large clinical trial underway examining the ability of allopurinol to prevent early renal loss. Several mechanisms have been proposed to explain the lower levels of SUA in type 1 diabetes including glucosuria induced uricosuria leading to spilling of urine uric acid (UUA) and lowering of SUA, and the notion that intracellular uric acid (IUA) and/ or UUA rather than SUA may be responsible for the development of complications. Animal studies have demonstrated that blocking uric acid production protects the kidney from tubulointerstitial injury, which suggests a causal role for uric acid in the development of diabetic tubular injury. Relative dehydration, secondary to glucosuria, exercise or inadequate liquid intake, may lead to concentrated and acidic urine, which may cause UUA to precipitate and crystallize in type 1 diabetes. The UUA precipitation and crystallization is thought to induce inflammation and injury of the tubules with possible retrograde glomerular injury. Moreover, it was recently shown that UUA promoted apoptosis in human proximal tubular cells by oxidative stress and activation of NADPH Oxidase NOX 4.

Oral alkali replacements are readily available, safe and include the following formulations sodium bicarbonate, BiCitra (sodium citrate and citric acid), PolyCitra (citric acid, sodium citrate, and potassium citrate), polycitra-K (potassium citrate and citric acid). In contrast to sodium bicarbonate, citrate is converted to bicarbonate in the liver and thus this conversion is affected by liver disease. Usual adult doses for urinary alkalinization are 325 to 2000 mg orally 1 to 4 times a day. One gram provides 12 mEq (mmoL) each of sodium and bicarbonate, and is titrated to a goal of urine pH of 8.0. In a prospective open-label trial 4 g of sodium bicarbonate was administered orally 3 times daily to 9 healthy volunteers for 24 hours, and after 10 hours all participants had a urine pH ≥ 7 and after 20 hours all participants had urine pH ≥ 8. No adverse effects or abnormal blood results were documented during the 24-hour follow-up. Urinary alkalinization should solubilize UUA thereby increasing the concentration of uric acid in urine and decreasing precipitation and crystallization of UUA. It is unknown whether alkalinization of urine reduces UUA precipitation and crystallization in type 1 diabetes.

With diabetic nephropathy being the leading cause of end-stage renal disease in the Western world, it is critical to develop a better understanding of the determinants of risk and progression of early diabetic nephropathy, to improve outcomes in patients with type 1 diabetes. UUA is a particularly attractive therapeutic target due to the potential to reduce tubular injury with sodium bicarbonate. Accordingly, the investigators propose a pilot experimental study examining the effect of urine alkalinization with oral sodium bicarbonate on UUA precipitation and crystallization in adults with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18-45 years) with type 1 diabetes
* Participants must be able to be fasting prior to study visit and give informed consent.

Exclusion Criteria:

* Non-type 1 diabetes
* History of eGFR <60 ml/min/1.73m2 or microalbuminuria or greater
* History of hypocalcemia or at risk of hypocalcemia
* Taking allopurinol or uric acid altering medications
* Ketogenic diet
* Ketonuria
* Taking phosphorus binders (e.g. sevelamer)
* Pregnant or breastfeeding
* Taking the following medications which may interact with sodium bicarbonate (e.g. phentermine, pseudoephedrine, antifungal medication, cephalosporin antibiotics [e.g. Keflex], tetracycline antibiotics [e.g. doxycycline], steroids or lithium)
* Taking SGLT-2 inhibitors
* Taking blood pressure medications

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-01; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Barbara Davis Center for Diabetes, Aurora, Colorado, United States

REFERENCES:
- [Background] Drummond K, Mauer M; International Diabetic Nephropathy Study Group. The early natural history of nephropathy in type 1 diabetes: II. Early renal structural changes in type 1 diabetes. Diabetes. 2002 May;51(5):1580-7. doi: 10.2337/diabetes.51.5.1580. PMID 11978659
- [Background] Gilbert RE, Cooper ME. The tubulointerstitium in progressive diabetic kidney disease: more than an aftermath of glomerular injury? Kidney Int. 1999 Nov;56(5):1627-37. doi: 10.1046/j.1523-1755.1999.00721.x. PMID 10571771
- [Background] Ginevri F, Piccotti E, Alinovi R, DeToni T, Biagini C, Chiggeri GM, Gusmano R. Reversible tubular proteinuria precedes microalbuminuria and correlates with the metabolic status in diabetic children. Pediatr Nephrol. 1993 Feb;7(1):23-6. doi: 10.1007/BF00861555. PMID 8439475
- [Background] Bjornstad P, Snell-Bergeon JK, McFann K, Wadwa RP, Rewers M, Rivard CJ, Jalal D, Chonchol MB, Johnson RJ, Maahs DM. Serum uric acid and insulin sensitivity in adolescents and adults with and without type 1 diabetes. J Diabetes Complications. 2014 May-Jun;28(3):298-304. doi: 10.1016/j.jdiacomp.2013.12.007. Epub 2013 Dec 27. PMID 24461546
- [Background] Bjornstad P, Lanaspa MA, Ishimoto T, Kosugi T, Kume S, Jalal D, Maahs DM, Snell-Bergeon JK, Johnson RJ, Nakagawa T. Fructose and uric acid in diabetic nephropathy. Diabetologia. 2015 Sep;58(9):1993-2002. doi: 10.1007/s00125-015-3650-4. Epub 2015 Jun 7. PMID 26049401
- [Background] Bjornstad P, Maahs DM, Rivard CJ, Pyle L, Rewers M, Johnson RJ, Snell-Bergeon JK. Serum uric acid predicts vascular complications in adults with type 1 diabetes: the coronary artery calcification in type 1 diabetes study. Acta Diabetol. 2014 Oct;51(5):783-91. doi: 10.1007/s00592-014-0611-1. Epub 2014 Jun 15. PMID 24929955
- [Background] Maahs DM, Caramori L, Cherney DZ, Galecki AT, Gao C, Jalal D, Perkins BA, Pop-Busui R, Rossing P, Mauer M, Doria A; PERL Consortium. Uric acid lowering to prevent kidney function loss in diabetes: the preventing early renal function loss (PERL) allopurinol study. Curr Diab Rep. 2013 Aug;13(4):550-9. doi: 10.1007/s11892-013-0381-0. PMID 23649945
- [Background] Lytvyn Y, Skrtic M, Yang GK, Yip PM, Perkins BA, Cherney DZ. Glycosuria-mediated urinary uric acid excretion in patients with uncomplicated type 1 diabetes mellitus. Am J Physiol Renal Physiol. 2015 Jan 15;308(2):F77-83. doi: 10.1152/ajprenal.00555.2014. Epub 2014 Nov 5. PMID 25377916
- [Background] Schepers MS, van Ballegooijen ES, Bangma CH, Verkoelen CF. Crystals cause acute necrotic cell death in renal proximal tubule cells, but not in collecting tubule cells. Kidney Int. 2005 Oct;68(4):1543-53. doi: 10.1111/j.1523-1755.2005.00566.x. PMID 16164631
- [Background] Ryu ES, Kim MJ, Shin HS, Jang YH, Choi HS, Jo I, Johnson RJ, Kang DH. Uric acid-induced phenotypic transition of renal tubular cells as a novel mechanism of chronic kidney disease. Am J Physiol Renal Physiol. 2013 Mar 1;304(5):F471-80. doi: 10.1152/ajprenal.00560.2012. Epub 2013 Jan 2. PMID 23283992
- [Background] Verzola D, Ratto E, Villaggio B, Parodi EL, Pontremoli R, Garibotto G, Viazzi F. Uric acid promotes apoptosis in human proximal tubule cells by oxidative stress and the activation of NADPH oxidase NOX 4. PLoS One. 2014 Dec 16;9(12):e115210. doi: 10.1371/journal.pone.0115210. eCollection 2014. PMID 25514209
- [Background] Cohen B, Laish I, Brosh-Nissimov T, Hoffman A, Katz LH, Braunstein R, Sagi R, Michael G. Efficacy of urine alkalinization by oral administration of sodium bicarbonate: a prospective open-label trial. Am J Emerg Med. 2013 Dec;31(12):1703-6. doi: 10.1016/j.ajem.2013.08.031. Epub 2013 Sep 20. PMID 24055481

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sodium Bicarbonate
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sodium Bicarbonate
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Type 1 Diabetes Duration [Mean (Standard Deviation); unit: years] | 20.2 (9.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Urine Uric Acid Concentration (Increased Solubility) by Assay
Description: Urine uric acid were evaluated using a QuantiChrom UA kit assay (DIUA-250) with quantitative colorimetric UA determination at 590 nm (BioAssay System, California, USA).
Time Frame: Day 1 (pre-therapy) and Day 2 (post-therapy)
Measure: Geometric Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Sodium Bicarbonate
Number analyzed (Participants) | 45
mg/dl
  Day 1 (pre-therapy) | 23.81 [18.93 to 29.94]
  Day 2 (post-therapy) | 22.30 [17.63 to 28.20]

2. Primary Outcome: Change in Number of Participants With Urine Uric Acid Precipitation by Polarized Microscopy
Description: Urine uric acid crystals were identified by polarized microscopy (Polarized light imaging Zeiss Axiovert 135; 0.3NA objective), and pictures were captured from each urine sample. UA crystals were defined dichotomously as being present or absent.
Time Frame: Day 1 (pre-therapy) and Day 2 (post-therapy)
Measure: Number; unit: participants
Arm/Group | Sodium Bicarbonate
Number analyzed (Participants) | 45
participants
  Day 1 (pre-therapy) | 14
  Day 2 (post-therapy) | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected while the participant was in the trial (24-36 hours)
Arm/Group | Sodium Bicarbonate
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 1/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sodium Bicarbonate (N=45)
Hypoglycemia (Endocrine disorders) | 1 (1) — Patient asked to fast and had a low serum blood glucose (31 mg/dl) with a normal point of care glucose (90 mg/dl) in clinic. Patient contacted upon receipt of serum glucose results. Patient asymptomatic with a normal glucose at the time of call.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT02502071/Prot_SAP_000.pdf